CLINICAL TRIAL: NCT06024785
Title: Comparison of Ligamentous Fixation Technique (Vertebropexy) Versus Conventional Decompression or Fusion Surgery for Degenerative Lumbar Spinal Disease: A Randomized Controlled Trial
Brief Title: Vertebropexy - Randomized-controlled Trial
Acronym: VPRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VPRCT
Record Dates: First submitted 2023-08-14; First posted 2023-09-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-11

CONDITIONS: Degeneration; Spinal Stenosis; Fusion of Spine
Keywords: degenerative lumbar spinal disease; decompression; fusion; vertebropexy; ligamentous fixation
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Intervention Model Description: * Stratification: Indication for decompression (study arm 1) or fusion (study arm 2)
  * Randomization within study arm 1 and study arm 2 between study intervention and control intervention
Masking Description: There is no blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Indication for decompression, randomization for decompression (Active Comparator): microsurgical (i.e., the use of a microscope or magnifying glasses during decompression) lumbar laminotomy with partial removal of the medial facet joint by preserving the midline structures (supraspinous-interspinous ligament complex); approach: bilateral or ipsilateral with cross-over to the contralateral side
  Interventions: Procedure: Vertebropexy
- Indication for decompression, randomization for vertebropexy (Experimental): decompression (see above) and additional stabilization of the spine with a ligament (for instance semitendinosus donor allograft), which connect the postoprior structures (Proc. Spinosus and/or Lamina) of the vertebrae . Situation-related application of laminar bands or analogous suture material (for instance FiberTape, Arthrex, Naples or Nile Band, K2M, Virginia)
  Interventions: Procedure: Vertebropexy
- Indication for fusion, randomization for fusion (Active Comparator): decompression (see above) and posterolateral instrumented fusion (arthrodesis) with implantation of pedicle screws, titanium alloy rods across the level of listhesis, an intervertebral fusion device and local autograft as well as DBX (demineralized bone matrix) to improve bony fusion
  Interventions: Procedure: Vertebropexy
- Indication for fusion, randomization for vertebropexy (Experimental): decompression (see above) and additional stabilization of the spine with a ligament (for instance semitendinosus donor allograft), which connect the postoprior structures (Proc. Spinosus and/or Lamina) of the vertebrae . Situation-related application of laminar bands or analogous suture material (for instance FiberTape, Arthrex, Naples or Nile Band, K2M, Virginia)
  Interventions: Procedure: Vertebropexy

INTERVENTIONS:
Procedure: Vertebropexy — microsurgical (i.e., the use of a microscope or magnifying glasses during decompression) lumbar laminotomy with partial removal of the medial facet joint by preserving the midline structures (supraspinous-interspinous ligament complex); approach: bilateral or ipsilateral with cross-over to the contralateral side. Additional stabilization of the spine with a ligament (for instance semitendinosus donor allograft), which connect the postoprior structures (Proc. Spinosus and/or Lamina) of the vertebrae . Situation-related application of laminar bands or analogous suture material (for instance FiberTape, Arthrex, Naples or Nile Band, K2M, Virginia)
  Other Names: ligamentous fixation of the spine

SUMMARY:
To assess the need for additional fusion surgery versus the risk of a revision surgery in patients with degenerative lumbar spinal disease and to assess efficacy and risk of the ligamentous fixation technique (vertebropexy)

DETAILED DESCRIPTION:
The global share of people over the age of 65 years has been consistently on the rise over the past few decades, and is still projected to increase. The increasing life expectancy, overall advances in medical care and therefore, the higher average age of people seeking surgical treatment lead to increasing numbers of spine surgeries: Spinal fusion is one of the most frequently used surgical treatment modalities for spinal disorders with 7.6 million per year worldwide (EU: 700,000, USA: 450,000, CH: 9000) and provides stability by internal rigid fixation of the spine with screws, rods and bony fusion. Although producing reliable short-term results with rapid pain relief and positive effects on patient outcome, implant-related complications, painful pseudarthrosis (non-union of bone), screw loosening, and adjacent segment disease lead to one-third of patients requiring reoperation within 15 years. These complications might be evoked by altered biomechanics with redistribution of loads and subsequently increased stress at the bone-implant interface as well as long fusions leading to relevant, irreversible loss of motion. Therefore, a new treatment modality which reinforces bony spinal segments with ligaments, the so called "vertebropexy", was recently developed by Farshad et al. The goal is to achieve targeted stabilization of the spine by inserting ligamentous allografts to counteract instability, without immobilizing the segment. Furthermore, it might provide additional stabilization after decompression surgery and therefore reduce revision surgery rates due to instability in clinically relevant directions as flexion-extension or anterior shear stress. However, to become a broadly accepted surgical alternative to existing surgical techniques for degenerative lumbar spinal disease like dorsal fusion and spinal decompression surgery, the new technique must provide convincing long-term results superior to those of these established procedures which is the primary objective of this randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Single-level or two-level lumbar surgery needed
* Indication for decompression surgery in patients with spinal canal stenosis and additional stable degenerative listhesis (without facet joint effusion ≥ 2mm)
* Indication for fusion surgery in patients with spinal canal stenosis and additional unstable degenerative listhesis (facet joint effusion ≥ 2mm), in patients with foraminal stenosis and additional degenerative listhesis, and in patients with segment degeneration of the disc
* Understanding in German language

Exclusion criteria:

* Indication for decompression and/or fusion surgery in patients with solely disc herniation, fractures, lytic listhesis, tumor
* Patients undergoing revision surgery for infection
* Patients undergoing revision surgery on the same level if bony structures have been removed (e.g. prior laminectomy or midline decompression)
* Patients undergoing revision surgery in case of prior fusion surgery
* Inability to understand the study for linguistic or cognitive reasons
* Anticipated clinical follow-up of less than 6 weeks after inclusion
* Participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
ODI (Oswestry Disability Index) | 2 years postoperative
  To assess and compare the clinical outcome of patients with spinal canal stenosis or foraminal stenosis +/- degenerative listhesis with either vertebropexy, decompression or fusion surgery

SECONDARY OUTCOMES:
VAS (Visual Analogue Scale) | 2 years postoperative
  To assess and compare the clinical outcome of patients with spinal canal stenosis or foraminal stenosis +/- degenerative listhesis with either vertebropexy, decompression or fusion surgery. VAS scale 0-10, 10 meaning the highest pain score and 0 no pain at all.
SSM symptoms/function (Spinal Stenosis Measure) | 2 years postoperative
  To assess and compare the clinical outcome of patients with spinal canal stenosis or foraminal stenosis +/- degenerative listhesis with either vertebropexy, decompression or fusion surgery
SSM satisfaction (Spinal Stenosis Measure) | 2 years postoperative
  To assess and compare the clinical outcome of patients with spinal canal stenosis or foraminal stenosis +/- degenerative listhesis with either vertebropexy, decompression or fusion surgery
EQ-5D (European Quality of Life Five Dimension) | 2 years postoperative
  To assess and compare the clinical outcome of patients with spinal canal stenosis or foraminal stenosis +/- degenerative listhesis with either vertebropexy, decompression or fusion surgery
Revision surgery | 2 years postoperative
  surgery on same and/or on adjacent levels
Complications | 2 years postoperative
  * - intraoperative: lesion of nerve root, dural tear, lesion of vessels
  * - postoperative: surgical site infection, wound healing disorder, hematoma, paresis, material loosening (with fusion), material failure (with fusion), pseudarthrosis (with fusion), fracture, allograft tendon rupture (with vertebropexy)
  * - non-surgical: anesthesiological, cardiovascular, pulmonal, thromboembolic, death
Duration of surgery | Perioperative
  Duration of intervention in minutes
Length of hospital stay | Perioperative
  Duration of hospital stay in days
Intraoperative blood loss | Perioperative
  Blood loss intraoperative in ml
Use of analgesia | 2 years postoperative
  Intake of analgetics
Use of physical therapy | 2 years postoperative
  Necessity to undergo further physical therapy (for instance due to remaining pain or function deficit)

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
The investigators affirm and uphold the principle of the participant's right to privacy and that they shall comply with applicable privacy laws. Especially, anonymity of the participants shall be guaranteed when presenting the data at scientific meetings or publishing them in scientific journals.
  Individual subject medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited. Subject confidentiality will be further ensured by utilising subject identification code numbers to correspond to treatment data in the computer files.
  For data verification purposes, authorised representatives of the Sponsor (-Investigator), a competent authority (e.g. Swissmedic), or an ethics committee may require direct access to parts of the medical records relevant to the study, including participants' medical history.

REFERENCES:
- [Background] Widmer J, Cornaz F, Scheibler G, Spirig JM, Snedeker JG, Farshad M. Biomechanical contribution of spinal structures to stability of the lumbar spine-novel biomechanical insights. Spine J. 2020 Oct;20(10):1705-1716. doi: 10.1016/j.spinee.2020.05.541. Epub 2020 May 28. PMID 32474224
- [Background] Farshad M, Tsagkaris C, Widmer J, Fasser MR, Cornaz F, Calek AK. Vertebropexy as a semi-rigid ligamentous alternative to lumbar spinal fusion. Eur Spine J. 2023 May;32(5):1695-1703. doi: 10.1007/s00586-023-07647-y. Epub 2023 Mar 17. PMID 36930387
- [Background] Calek AK, Widmer J, Fasser MR, Farshad M. Lumbar vertebropexy after unilateral total facetectomy. Spine J. 2023 Nov;23(11):1730-1737. doi: 10.1016/j.spinee.2023.07.005. Epub 2023 Jul 13. PMID 37451550
- [Background] Calek AK, Altorfer F, Fasser MR, Widmer J, Farshad M. Interspinous and spinolaminar synthetic vertebropexy of the lumbar spine. Eur Spine J. 2023 Sep;32(9):3183-3191. doi: 10.1007/s00586-023-07798-y. Epub 2023 Jun 7. PMID 37284900